CLINICAL TRIAL: NCT01701011
Title: Study of the Effectiveness of a Coping Selfhelp Intervention for Women in the Waiting Period After an Embryo Transfer During an IVF/ISCI Treatment
Brief Title: Coping Intervention After Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bart CJM Fauser (Other)
Responsible Party: Sponsor-Investigator, Bart CJM Fauser, prof, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: PRCI study
Record Dates: First submitted 2010-10-06; First posted 2012-10-04 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-06

CONDITIONS: Anxiety; Depression
Keywords: coping; intervention; waiting-period
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PRCI-monitoring (Experimental): Coping intervention, Daily Record Keeping, Questionnaires
  Interventions: Behavioral: Coping intervention
- Routine care control (No Intervention): Questionnaires
- Monitoring control (No Intervention): DRK and Questionnaires

INTERVENTIONS:
Behavioral: Coping intervention — Positive reappraisal coping intervention
  Arms: PRCI-monitoring

SUMMARY:
Background of the study:

Undergoing an IVF or ICSI treatment is an emotional and physical burden for both the woman and her partner. Most stressful for the couple is waiting for the result of the treatment, the period after the embryotransfer until the pregnancy test or menstruation and an unsuccessful treatment. Symptoms of anxiety and depression have been identified in couples during the waitingperiod after an embryotransfer. For this waitingperiod a short selfhelp copingintervention has been developed based on the stress theory of Lazarus for women to use at home. Goal of the instrument is to stimulate the copingstyle positive reappraisal. Research has demonstrated that using this copingstyle can have a positive impact in health related circumstances.

DETAILED DESCRIPTION:
Objective of the study:

To investigate if a short copingintervention reduces anxiety in patients undergoing an IVF or ICSI treatment in the UMCU during the waitingperiod after an embryotransfer.

Study design:

In this research a randomised controlled trial (RCT) will be used for three groups. The choice for three groups has been based on earlier research with a daily record keeping (DRK). The DRK is a daily measurement for emotions, copingstyle and physical complaints. Previous research with the DRK showed an increase of anxiety. More research must be done of the impact of the DRK. Group 1: Positive Reappraisal Coping Intervention (PRCI) & DRK & questionnaires Group 2: DRK & questionnaires Group 3: Standard care & questionnaires

Study population:

Patients undergoing an IVF or ICSI treatment in the UMCU.

Intervention (if applicable):

A selfhelp coping intervention

Primary study parameters/outcome of the study:

Anxiety

Secondary study parameters/outcome of the study (if applicable):

Risk of emotional problems copingstyle depression vital pregnancy quality of life

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable):

Using the coping intervention may reduce anxiety for the patient. The use of this instrument is not a burden for patients. The burden for patients is to complete questionnaires before, during and six weeks after the embryotransfer. Partners are asked to fill in a questionnaire at three times.

ELIGIBILITY:
Inclusion Criteria:

* Patient in IVF/ICSI treatment

Exclusion Criteria:

* Patient who do not speak the dutch language

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: N.S. Macklon, MD, PhD, Principal Investigator — University of Southampton; J Boivin, PhD, Principal Investigator — Cardiff University
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Ockhuijsen H, van den Hoogen A, Eijkemans M, Macklon N, Boivin J. The impact of a self-administered coping intervention on emotional well-being in women awaiting the outcome of IVF treatment: a randomized controlled trial. Hum Reprod. 2014 Jul;29(7):1459-70. doi: 10.1093/humrep/deu093. Epub 2014 May 7. PMID 24812317
- [Derived] Ockhuijsen HD, van den Hoogen A, Macklon NS, Boivin J. The PRCI study: design of a randomized clinical trial to evaluate a coping intervention for medical waiting periods used by women undergoing a fertility treatment. BMC Womens Health. 2013 Sep 3;13:35. doi: 10.1186/1472-6874-13-35. PMID 24004640
- See also: Article study protocol — http://www.biomedcentral.com/content/pdf/1472-6874-13-35.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the 20 months of recruitment, between October 2010 and June 2012, 1445 letters were sent to women with an invitation to the trial.
Pre-assignment Details: Of the 565 women who replied via a letter or email, 188 (33%) were not eligible. The remaining 377 women were randomised and the 349 who had an embryo to transfer (n=119 PRCI-monitoring, n=117 monitoring-control, n=113 routine care control)
Groups:
- PRCI-monitoring Group: Coping intervention, Daily Record Keeping, Questionnaires
- Monitoring-control Group: Daily Record Keeping and Questionnaires
- Routine Care Control Group: Patients receive only questionnaires
Period: Overall Study
Arm/Group | PRCI-monitoring Group | Monitoring-control Group | Routine Care Control Group
Started | 127 | 126 | 124
Completed | 92 | 102 | 90
Not Completed | 35 | 24 | 34

BASELINE CHARACTERISTICS:
Groups:
- PRCI-monitoring Group: Coping intervention, Daily Record Keeping, Questionnaires
  Coping intervention, Daily Record Keeping, Questionnaires :
- Monitoring-control Group: DRK and Questionnaires
  Coping intervention, Daily Record Keeping, Questionnaires :
- Routine Care Control Group: Questionnaires
  Coping intervention, Daily Record Keeping, Questionnaires :
- Total: Total of all reporting groups
Arm/Group | PRCI-monitoring Group | Monitoring-control Group | Routine Care Control Group | Total
Number analyzed (Participants) | 127 | 126 | 124 | 377
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (4.7) | 34.6 (4.7) | 34.8 (5.0) | 34.8 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 126 | 124 | 377
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 127 | 126 | 124 | 377

OUTCOME MEASURES:

1. Primary Outcome: Anxiety
Description: The Hospital Anxiety and Depression Scale (HADS) was used to measure general anxiety and depression (Zigmond and Snaith, 1983). TheHADSconsists of 14 items (7 items for each subscale) that are rated on a 4-point Likert scale. The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0 to 21). Scores on each scale can be interpreted in ranges: normal (0-7), mild (8-10), moderate (11-14) and severe (15-21) anxiety and depression.
Time Frame: T1 during the first week of the stimulation phase, T2 on the 10th day after embryo transfer, T3 six weeks after embryo transfer
Population: Only in women with embryo transfer
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Routine Care Control Group: patients receive questionnaires
Arm/Group | PRCI-monitoring Group | Monitoring-control Group | Routine Care Control Group
Number analyzed (Participants) | 119 | 117 | 113
units on a scale
  Time 1 | 6.279 (0.242) | 6.223 (0.243) | 6.095 (0.251)
  Time 2 | 7.302 (0.269) | 7.526 (0.249) | 8.175 (0.272)
  Time 3 | 5.798 (0.279) | 5.571 (0.262) | 6.317 (0.288)
Statistical Analysis 1: Comparison: Monitoring-control Group vs Routine Care Control Group; IBM SPSS Statistics 20 was used to perform the statistical analysis. A mixed model for repeated measures was used to examine the differences between the three groups over time for the primary outcome, anxiety. All models were estimated by the method of restricted maximum likelihood (REML) and the Compound Symmetry covariance structure was chosen for the repeated measures. The analysiswas performed according to the intention to treat; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: PRCI-monitoring Group vs Monitoring-control Group vs Routine Care Control Group; To test the difference in psychological well-being between three groups with a power of 95%,a ¼ 0.05 and a medium effect size ( f ¼ 0.25), a total of 297 participants were required (99 patients per group). Taking into account a 20% attrition rate, at least 124 women had to be recruited in each group; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Depression
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Only in women with embryo transfer
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | PRCI-monitoring Group | Monitoring-control Group | Routine Care Control Group
Number analyzed (Participants) | 119 | 117 | 113
units on a scale
  Time 1 | 3.389 (0.199) | 3.391 (0.201) | 3.269 (0.208)
  Time 2 | 3.709 (0.222) | 3.676 (0.206) | 4.224 (0.225)
  Time 3 | 3.983 (0.230) | 3.708 (0.216) | 3.736 (0.238)
Statistical Analysis 1: Comparison: Monitoring-control Group vs Routine Care Control Group; IBM SPSS Statistics 20 was used to perform the statistical analysis. A mixed model for repeated measures was used to examine the differences between the three groups over time for the secondary outcome, depression. All models were estimated by the method of restricted maximum likelihood (REML) and the Compound Symmetry covariance structure was chosen for the repeated measures. The analysiswas performed according to the intention to treat; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Groups:
- Routine Care Control Group: patients received questionnaires
Arm/Group | PRCI-monitoring Group | Monitoring-control Group | Routine Care Control Group
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/126 | 0/124
Other Adverse Events (participants affected / at risk) | 0/127 | 0/126 | 0/124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes